CLINICAL TRIAL: NCT03078231
Title: Pilot Assessment of EyeArt as an Automated Diabetic Retinopathy Screening Tool
Status: Completed | Type: Observational
Sponsor: Eyenuk, Inc. (Industry)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: EN-01p; 9SB1EY027241 (NIH); 2R44EY026864 (NIH)
Record Dates: First submitted 2017-03-02; First posted 2017-03-13 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Mydriatics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

INTERVENTIONS:
Procedure: Color fundus photography — Subjects will undergo fundus photography before and after administration of mydriatic agent.
Drug: Mydriatic Agent — Subjects will be administered mydriatic medication to dilate their pupils.

SUMMARY:
More than 29 million people in the US are living with diabetes, many of whom will develop diabetic retinopathy (DR) or diabetic eye disease (DED), the leading cause of vision loss and blindness in working-age adults. Annual eye screening is recommended for all diabetic patients since vision loss can be prevented with laser photocoagulation and anti-VEGF injections if DR is diagnosed in its early stages. Currently, the number of clinical personnel trained for DR screening is orders of magnitude smaller than that needed to screen the large, growing diabetic population. Therefore, to meet this large unmet need for DR screening, a fully-automated computerized DR screening system is necessary. This study is designed to assess the performance of EyeArt, an automated DR screening tool.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* a diagnosis of diabetes mellitus; and
* understanding of study and provision of written informed consent.

Exclusion Criteria:

* Persistent visual impairment or sudden vision loss in one or both eyes;
* History of uncorrected media opacity in one or both eyes;
* History of retinal vascular disease other than diabetic eye disease;
* History of ocular injections, laser treatment of the retina, or intraocular surgery other than cataract;
* Subject has contraindications for mydriatic medications or is unwilling or unable to dilate;
* Subject is currently enrolled in an interventional study of an investigational device/drug; or
* Subject has a condition or is in a situation which in the opinion of the Investigator, might confound study results, may interfere significantly with the subject's participation in the study, or result in ungradable 4-wide field stereoscopic mydriatic fundus photographs.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study subjects will be enrolled at a primary care center
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2017-04-24 (Actual); Study Completion 2017-04-24 (Actual)

PRIMARY OUTCOMES:
Number of subjects whose EyeArt results match the reading center grading for identifying referable diabetic eye disease (moderate NPDR or higher on the ICDR scale or surrogate markers for CSME). | 1 visit
  The performance of EyeArt will be evaluated using overall accuracy, sensitivity, and specificity measures.

CONTACTS AND LOCATIONS:
Locations (1):
- LAC+USC Medical Center, Los Angeles, California, United States